CLINICAL TRIAL: NCT01496443
Title: A Phase 1, Single-Blind, Placebo Controlled, Sequential Design Study to Evaluate the Drug Interaction Potential Between Glimepiride and TAK-875 in Subjects With Type 2 Diabetes Mellitus
Brief Title: TAK-875 Glimepiride Drug-Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: TAK-875_118; U1111-1126-0128 (Registry Identifier: WHO)
Record Dates: First submitted 2011-12-18; First posted 2011-12-21 (Estimated); Last update posted 2012-09-13 (Estimated); Status verified 2012-09

CONDITIONS: Pharmacokinetics
Keywords: Drug Therapy
MeSH Terms: interventions — TAK-875; glimepiride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- TAK-875 & Glimepiride QD (Experimental): TAK-875 50 mg, tablets, orally and glimepiride 2 mg, capsules, orally and glimepiride placebo matching capsules, orally, once daily on dosing days for up to 19 days.
  Interventions: Drug: TAK-875 and Glimepiride

INTERVENTIONS:
Drug: TAK-875 and Glimepiride
  Other Names: Amaryl

SUMMARY:
The purpose of this study is to determine the pharmacokinetics and safety of TAK-875, once daily (QD), with and without glimepiride in participants with type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
TAK-875 is being developed at Takeda Global Research and Development, Inc. as an adjunct to diet and exercise to improve glycemic control in participants with T2DM.

This study will determine whether administration of glimepiride alters the pharmacokinetics (PK) of TAK-875, and whether TAK-875 affects the PK of glimepiride.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. The participant is a male or female with T2DM who is newly diagnosed, managed with diet and exercise alone, or taking up to 2 oral antidiabetic agents (except insulin and thiazolidinediones (TZDs)) and willing to discontinue the antidiabetic medications 2 weeks prior to enrollment.
4. The participant is aged 18 to 68 years, inclusive, at the time of informed consent and on Day 1.
5. The participant weighs at least 50 kg (110 lb) and has a body mass index (BMI) between 18.0 and 40.0 kg/m2, inclusive at Screening.
6. A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 30 days after last dose.
7. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent throughout the duration of the study and for 30 days after last dose.
8. The participant has an fasting serum glucose (FPG) >126 mg/dL and <260 mg/dL if not on any diabetic medication, or <220 mg/dL if on any single antidiabetic agent, or < 200 mg/dL if on any combination of 2 oral antidiabetic agents at Screening.
9. The participant has a fasting C-peptide concentration ≥0.8 ng/mL at Screening.
10. The participant has not received treatment with weight-loss drugs within the 3 months prior to Screening.
11. The participant has a systolic blood pressure ≤160 mmHg and a diastolic blood pressure of ≤100 mmHg at Screening and at Check-in (Day -1).
12. The participant met one of the following glycated hemoglobin (HbA1c) criteria (diagnosis must be based on current American Diabetes Association (ADA) criteria) at Screening:

    * Participant who is treatment naïve should have an HbA1c concentration ≥6.5% and ≤10.0%.
    * Participant who is on a single antidiabetic agent (stable dose for at least 28 days) should have an HbA1c ≥6% and ≤9.5%.
    * Participant who is on a combination of up to 2 antidiabetic agents (stable doses for at least 28 days) should have an HbA1c ≥6% and ≤9.0%.
13. The participant has negative test results at Screening and Check-in (Day -1) for selected substances of abuse including alcohol and cotinine.
14. The participant has Screening and Check-in (Day -1) clinical laboratory evaluations (including fasting clinical chemistry, hematology, and complete urinalysis [excluding glucose results]) within the reference range for the testing laboratory, unless the investigator deems the out-of-range results to be not clinically significant.
15. The participant is willing to refrain from strenuous exercise from 72 hours before Check-in (Day -1) and throughout study.
16. The participant is considered by the investigator to be in good health (other than being diabetic) as determined during the medical history review, physical examination findings, electrocardiogram (ECG) and vital sign results, and clinical laboratory evaluations.
17. The participant has a normal creatinine clearance of >60 mL/min using the Cockcroft-Gault formula at Screening and Check-in (Day -1).

Exclusion Criteria:

1. The participant is participating in another investigational study or has taken any investigational drug within 30 days prior to Check-in (Day -1).
2. The participant has received TAK-875 in a previous clinical study.
3. The participant's QTcF (Fridericia's correction) is >450 msec (for both male and female participants) at Screening or at Check-in (Day -1) as read on the printout of the ECG produced by the ECG equipment or manually calculated and then evaluated by the investigator.
4. The participant has a resting pulse or heart rate <45 bpm or >100 bpm at Screening or Check-in (Day -1).
5. The participant is an immediate family member, study site employee, or in a dependent relationship with a study site employee who is involved in the conduct of this study (e.g., spouse, parent, child, sibling) or may consent under duress.
6. The participant is on any insulin or TZD treatment.
7. Participant has a known hypersensitivity to any component of the formulation of TAK-875 or glimepiride (see Package Insert).
8. The participant has a positive urine drug result for drugs of abuse at Screening or Check-in (Day -1).
9. The participant has a history of proteinuria >300 mg/day on a 12- or 24-hour urine collection or an albumin/creatinine ratio >300 μg/mg at Screening. If elevated, the participant may be rescreened within 1 week, and may be included in study with agreement between Principal Investigator and the TGRD Medical Monitor.
10. The participant has a history of "severe" hypoglycemia (as defined in Section 7.5.1) within 4 weeks prior to Screening.
11. The participant has a history of any clinically significant retinopathy, which is defined as more than moderate nonproliferative diabetic retinopathy or any stage of proliferative diabetic retinopathy or any history of laser-treated retinopathy.
12. The participant has a history of treated or clinically significant peripheral or autonomic neuropathy.
13. The participant has a history of ulcerative colitis or Crohn's disease, or has undergone gastric resection.
14. The participant has a history of a psychiatric disorder that will affect the participant's ability to participate in the study.
15. The participant has a history of angioedema.
16. The participant had an acute, clinically significant illness within 30 days prior to Check-in (Day -1), or any other condition or prior therapy that, in the opinion of the investigator, would make the participant unsuitable for the study.
17. The participant has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse (defined as regular or daily consumption of more than 4 alcoholic drinks per day) within 1 year prior to the Screening visit or is unwilling to agree to abstain from alcohol and drugs throughout the study.
18. Participant has taken any excluded medication, supplements or food products.
19. If female, the participant is pregnant or lactating or intending to become pregnant before, during, or within 30 days after participating in this study; or intending to donate ova during such time period.
20. If male, the participant intends to donate sperm during the course of this study or for 30 days after the last dose of study drug.
21. The participant has a history of cardiac arrhythmia, systolic dysfunction congestive heart failure, angina, myocardial ischemia or infarction, or stroke within 1 year prior to Screening, or the presence of an abnormal ECG that, in the investigator's opinion, is clinically significant.
22. Participant has current or recent (within 6 months) gastrointestinal disease that would be expected to influence the absorption of drugs (i.e., a history of malabsorption, esophageal reflux, peptic ulcer disease, erosive esophagitis, frequent [more than once per week] occurrence of heartburn, or any surgical intervention [e.g., cholecystectomy]).
23. The participant has a total bilirubin >1.5 mg/dL at Screening or Check-in (Day -1).
24. Participant has abnormal Screening or Check-in (Day -1) laboratory values that suggest a clinically significant underlying disease or participant with the following lab abnormalities: ALT and/or Aspartate Aminotransferase (AST) level >2x ULN for the testing laboratory, active liver disease, or jaundice at Screening or Check-in (Day -1).
25. The participant has a history of abdominal surgery (except laparoscopic cholecystectomy or uncomplicated appendectomy), thoracic or nonperipheral vascular surgery within 6 months prior to Check-in (Day -1).
26. Participant has a history of cancer, other than basal cell or Stage 1 squamous carcinoma of the skin that has not been in remission for at least 5 years prior to Day 1.
27. Participant has a positive test result for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV), or a known history of human immunodeficiency virus infection at Screening.
28. Participant has used any nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patch or nicotine gum) within 28 days prior to Check-in (Day -1) or is unwilling to abstain from these products for the duration of the study or has a positive cotinine test result at Screening or Check-in (Day -1).
29. The participant has poor peripheral venous access.
30. The participant is unwilling or unable to comply with the protocol or scheduled appointments.
31. The participant is unable to understand verbal and/or written English or any other language for which a certified translation of the approved informed consent is available.
32. The participant has donated blood or experienced acute blood loss (including plasmapheresis) of >500 mL within 90 days prior to Day 1.
33. Participant has a Screening or Check-in (Day -1) abnormal (clinically significant) ECG. Entry of any participant with an abnormal (not clinically significant) ECG must be approved, and documented by signature of the principal investigator.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Cmax: Maximum Observed Plasma Concentration Pharmacokinetic Parameter for TAK-875 | Day 17 and Day 18.
  Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.
Cmax: Maximum Observed Plasma Concentration Pharmacokinetic Parameter for Glimepiride | Day 1 and Day 18.
  Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.
Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) Pharmacokinetic Parameter for TAK-875 | Day 17 and Day 18.
  Time to reach the maximum plasma concentration (Cmax), equal to time (hours) to Cmax.
Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) Pharmacokinetic Parameter for Glimepiride | Day 1 and Day 18.
  Time to reach the maximum plasma concentration (Cmax), equal to time (hours) to Cmax
AUC(0-tlqc): Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration Pharmacokinetic Parameter for Glimepiride | Day 1 and Day 18.
  (AUC(0-tlqc) is a measure of total plasma exposure to the drug from Time 0 to Time of the Last Quantifiable Concentration (AUC[0-tlqc]).
AUC(0-inf): Area Under the Plasma Concentration-time Curve from Time 0 to Infinity Pharmacokinetic Parameter for Glimepiride | Day 1 and Day 18.
  AUC(0-inf) is measure of area under the plasma concentration-time curve from time 0 to infinity after drug administration.
AUC(0-24): Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours Postdose Pharmacokinetic Parameter for TAK-875 | Day 17 and Day 18.
  AUC(0-24) is measure of area under the curve over the dosing interval (tau) (AUC(0-tau]), where tau is the length of the dosing interval - 24 hours in this study).

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Clinical Science, Study Director — Takeda
Locations (1):
- San Antonio, Texas, United States